CLINICAL TRIAL: NCT07243158
Title: A Prospective, Multicenter, Randomized Controlled Clinical Study to Evaluate the Safety and Effectiveness of the DragonFly Transcatheter Mitral Valve Clip System in the Treatment of Moderate-to-Severe or Severe Functional Mitral Regurgitation (FMR)
Brief Title: Randomized Controlled Study of Dragonfly System for Functional Mitral Regurgitation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Valgen Medtech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DragonFly-03
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Mitral Regurgitation Functional
MeSH Terms: interventions — Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Randomized - Device Group (Experimental): This group is allocated to use DragonFly System for edge-to-edge repair manufactured by Hangzhou Valgen Medtech Co., Ltd.
  Interventions: Device: DragonFly System; Drug: Drug
- Randomized - Control Group (Active Comparator): This group will continue to be managed on medical therapy, per physician discretion
  Interventions: Device: DragonFly System; Drug: Drug

INTERVENTIONS:
Device: DragonFly System — This group is allocated to use DragonFly System for edge-to-edge repair manufactured by Hangzhou Valgen Medtech Co., Ltd.
Drug: Drug — This group will continue to be managed on medical therapy, per physician discretion

SUMMARY:
To confirm the effectiveness and safety of the Dragonfly transcatheter mitral valve repair system for the treatment of chronic moderate to severe (3+) or severe (4+) functional mitral regurgitation (FMR) who remained clinically symptomatic after adequate treatment.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, randomized controlled design. Patients are chronic moderate to severe (3+) or severe (4+) functional mitral regurgitation (FMR) who remained clinically symptomatic after guideline-directed medical treatment. After signing an informed consent form, subjects in the experimental group will undergo the transcatheter mitral valve repair procedure using the DragonFly™ Transcatheter Mitral Valve Clip System . According to the investigator's discretion, all subjects in the treatment group will continue to receive maximally tolerated guideline-directed medical therapy (GDMT). Subjects in the control group will also continue maximally tolerated GDMT as determined by the investigator. After completing the 12-month follow-up, crossover to the treatment group will be permitted.

All subjects were followed up before discharge (excluding the control group), and 30 days, 6 months, 12 months, and 24 months after treatment. Subjects in the experimental group and those who crossed over to the experimental group underwent extended clinical follow-up for 3, 4, and 5 years.

ELIGIBILITY:
Inclusion Criteria:

1) Age ≥ 18 yrs. 2) Symptomatic functional mitral regurgitation (FMR) (≥3+) due to ischemic or non-ischemic cardiomyopathy

* Transseptal catheterization and femoral vein access is determined to be feasible.
* The subject or subject's legal representative has been informed of the nature of the trial, willing to accept the experimental tests, and has provided written informed consent.

Exclusion Criteria:

1) Echocardiographic evidence of intracardiac mass, thrombus, or vegetation. 2）Echocardiography revealed severe restriction of leaflet motion due to tethering.

3) The presence of other severe heart valve disease requiring surgical intervention.

* Currently participating in an investigational drug or another device study that has not completed its primary endpoints or would clinically interfere with the endpoint of this study. Note: Trials requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational trials.
* In the judgment of the investigator, subjects may not complete the trial according to poor compliance or in other circumstances when the investigator determines that the subject is unfit to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical success at 12 months after the procedure | 12 months
  The rate of the composite endpoint of freedom from all-cause mortality, hospitalization for heart failure, NYHA improved <1 class and MR > 2+ at 12 months.

SECONDARY OUTCOMES:
Mitral regurgitation severity | 30 days, 6 months, 12 months
  Percentage of patients with mitral regurgitation of 2+ or less.
Recurrent heart failure (HF) hospitalizations | 30 days, 6 months, 12 months
  Number of patients with incidence of re-hospitalizations for heart failure after Dragonfly implantation.
NYHA Class | 30 days, 6 months, and 12 months
  Number of patients with New York Heart Association (NYHA) Function Class I or II.
Change in 6 minutes walk test distance | 12 months
  Improvement in 6 Minute Walk Test distance at 12 months over baseline.
Quality of life improvement | 12 months
  Improvement in quality of life (QoL) at 12 months over baseline, as measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ).
Left Ventricular End Diastolic Volume (LVEDV) | 12 months
  Left Ventricular End Diastolic Volume (LVEDV) as determined by the core echocardiography laboratory from a transthoracic echocardiogram (TTE).
Acute procedural success（only for experimental group） | Immediately after procedure, Discharge: The day after the patient's exit from the cardiac catheterization laboratory
  Successful in Dragonfly implantation, and residual MR of 2+ or less at discharge. An echocardiography echocardiogram at 30 days can be accepted if the discharge image was not available or hard to interpret. A death before discharge or a re-operation of mitral valve prior to 30 days is defined as acute procedure failure.
Acute device success（only for experimental group） | Immediately after procedure
  One or more Dragonfly devices are successfully delivered and released, edge-to-edge leaflet repair confirmed by echocardiogram, and successfully withdrawal of the delivery catheter.

OTHER OUTCOMES:
Incidence of adverse events | 12 months
  MAE is defined as a combined clinical endpoint of single leaflet device attachment (SLDA), device embolization, endocarditis requiring surgery, mitral stenosis confirmed by the echocardiographic core laboratory requiring surgical intervention, left ventricular assist device (LVAD) implantation, heart transplantation, and nonelective cardiovascular surgery for device or procedure-related adverse events occurring after transseptal catheterization.（only for experimental group）
Incidence of major adverse events (MAEs) | 30 Days
  MAE is defined as a combined clinical endpoint of death, stroke, myocardial infarction, and nonelective cardiovascular surgery for device or procedure-related adverse events occurring after transseptal catheterization.（only for experimental group）
All-cause mortality | 12 months
  Percentage of all-cause death includes cardiac death, non-cardiac death, and death from unknown causes.

CONTACTS AND LOCATIONS:
Overall Officials: Jianan Wang, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No